CLINICAL TRIAL: NCT01413217
Title: "Which is a Better Breakfast? Egg or Cereal?"
Brief Title: Which is a Better Breakfast? Egg or Cereal?
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: American Egg Board (Other)
Responsible Party: Sponsor
Other Study IDs: PBRC 10010
Record Dates: First submitted 2011-07-15; First posted 2011-08-10 (Estimated); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Hunger; Satiety

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Egg Breakfast: This group will be given a breakfast consisting of eggs. A breakfast consisting of eggs induces greater satiety and reduces Lunch Time intake.
- Cereal Breakfast: This breakfast will consist of a breakfast that will include cereal. A breakfast cereal or white bread increases lunchtime energy intake.

SUMMARY:
Which is a better breakfast? Egg or cereal?

DETAILED DESCRIPTION:
Which breakfast has the most beneficial effect on blood glucose and insulin, blood hormones and blood pressure, egg or cereal breakfast? Over a seven week period the participant will take part in eating breakfast of either egg breakfast or cereal breakfast which will be monitored. Blood samples will be taken before participants eat and different times throughout until after Lunch on day 1 and day 7. Questionnaires will be given to determine satiety (feeling of fullness) and hunger before and after breakfast and lunch. After a two week period participants will return for another week of the same procedure and tests that was followed from Day 1 though day 7 listed. However, this time participants will be eating the second of the two breakfasts whichever one they did not have for the first test period.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age
* not lost more than 5% of body wight in the past 3 months, or not trying to actively lose weight at the moment.
* are not suffering from disease such as major heart conditions, cancer, type 1 diabetes, eating disorders, very high cholesterol or triglycerides levels, or any serious illness that requires intensive and long term medical treatment.

are not allergic to or sensitive to eggs, soy or wheat, and do not dislike these foods.

* have a BMI of equal to or >30 to equal to or <60

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In the community area of Baton Rouge, LA area exclusively random process to guarantee that each participant or population has specified chance of selection.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Caloric intake for Lunch after you have received an Egg or Cereal Breakfast and Levels of glucose, insulin, and lipids are measured. | 7 weeks
  Before breakfast satiety following an egg breakfast compared to the other breakfast determines the impact of egg breakfast on their Lunch intake. Blood samples will be taken to test the levels of glucose, insulin, and lipids like cholesterol and triglycerides.

SECONDARY OUTCOMES:
Satiety or hunger | 7 weeks
  Questionnaires to determine satiety and/or hunger before and after breakfast and lunch will be given.

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Bayham BE, Greenway FL, Johnson WD, Dhurandhar NV. A randomized trial to manipulate the quality instead of quantity of dietary proteins to influence the markers of satiety. J Diabetes Complications. 2014 Jul-Aug;28(4):547-52. doi: 10.1016/j.jdiacomp.2014.02.002. Epub 2014 Feb 13. PMID 24703415